CLINICAL TRIAL: NCT05376865
Title: The Interactive Effect of Vitamin D3 Supplementation and Vitamin D Receptor Polymorphisms on Obesity, Inflammatory and Metabolic Markers in Overweight Women With Hypovitaminosis D
Brief Title: Effects of Vitamin D Supplementation on Obesity, Inflammatory and Metabolic Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tirang R. Neyestani, Ph.D. (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Tirang R. Neyestani, Ph.D., Prof., National Nutrition and Food Technology Institute
Organization: National Nutrition and Food Technology Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Overweight; Hypovitaminosis D
MeSH Terms: conditions — Overweight; Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Vitamin D3 supplement every week
  Interventions: Dietary Supplement: Vitamin D supplement
- Control (Placebo Comparator): Placebo every week
  Interventions: Dietary Supplement: Vitamin D supplement

INTERVENTIONS:
Dietary Supplement: Vitamin D supplement — The intervention group receives 50000 IU of vitamin D every week as vitamin D supplements for 12 weeks, provided monthly.

SUMMARY:
46 eligible overweight women with hypovitaminosis D are assigned to either vitamin D or control group using block randomization method. Vitamin D3 pearl (Zahravi Pharma Co, Tabriz, Iran) containing 50000 IU cholecalciferol or placebo are administered weekly for 12 weeks. Participants in both groups are structured to hold their sun exposure and physical activity habits and not take any vitamin supplements during the study.

DETAILED DESCRIPTION:
For the randomized controlled clinical trial (RCT), the first fifty eligible women were assigned to either the vitamin D or placebo group using the block randomization method. Each Vitamin D3 pearl (Zahravi Pharma Co, Tabriz, Iran) contained 50000 IU cholecalciferol and was administered weekly for 12 weeks according to guidelines for treating vitamin D deficiency. Placebo pearls (Zahravi Pharma Co, Tabriz, Iran) had the identical appearance, taste, and smell as the vitamin D pearls and could only be identified by the package code. The placebo pearls were administered similarly. To keep the study double-blinded, an assistant who was not involved in assessments managed the randomization and supplement assignment procedure. Participants were structured to hold their sun exposure and physical activity habits and not take any vitamin supplements during the study. They were also asked to inform the researcher before taking any new medications. All participants were provided with a moderately reduced diet (a reduction of 300 kcal per day) based on their basal weight. The nutrigenetic study investigated 75 eligible women (including the vitamin D group and the last fifty women who entered the study). The nutrigenetic study protocol was the same as that mentioned above for the vitamin D group in the RCT. Compliance was ensured by weekly text messages and voice calls to remind the users of the supplement on the given day. In addition, the supplement and placebo pearls were presented in two visits; once at the baseline visit and then after six weeks. Pearls packs were collected from each subject (at week 6 and week 12) to check if all the pearls were consumed as recommended.

During the first and last visits, anthropometric and laboratory assessments were performed for all subjects. The primary outcomes are improving anthropometric, inflammatory, and metabolic markers of overweight women with hypovitaminosis D.

ELIGIBILITY:
Inclusion Criteria:

* low serum vitamin D level <30ng/ml
* 25<BMI<30 kg/m2
* Age: 20-50
* Free of chronic diseased such as cancer, diabetes, cardiovascular disease, renal diseases, gastrointestinal diseases, no multivitamin supplement intake, no change in weight in the last 3 months

Exclusion Criteria:

* Getting pregnant during the study
* Suffering from thyroid disorders and other diseases mentioned during the study
* Not taking supplements weekly

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Serum 25(OH)D | 12 weeks
  Fasting serum 25-hydroxyvitamin D level
Weight | 12 weeks
  Subject's weight wearing light clothing

SECONDARY OUTCOMES:
Waist circumference | 12 weeks
  the measurement at the midpoint between the lowest rib and the iliac crest
Fat mass | 12 weeks
  Total body fat mass measured by Bioelectrical Impedance analysis method
Serum Fasting Glucose | 12 weeks
  Fasting serum glucose level
Serum total cholesterol | 12 weeks
  Fasting serum total cholesterol level
Serum triglyceride | 12 weeks
  Fasting serum triglyceride level Fasting serum triglyceride leve
Serum hsCRP | 12 weeks
  Fasting serum high sensitivity c-reactive protein level
Serum IL-6 | 12 weeks
  Fasting serum Interleukin-6 level
Serum TNF-a | 12 weeks
  Fasting serum tumor necrosis factor alpha level
Serum PTH | 12 weeks
  Fasting serum parathyroid hormone level

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Nutrition Research, National Nutrition and Food Technology Research Institute (NNFTRI) and Faculty of Nutrition Science and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran, Tehran, Iran